CLINICAL TRIAL: NCT07056088
Title: A Randomized Controlled Trial Comparing Blood Glucose Control Intraoperative Between Insulin Drip vs. Insulin Boluses
Brief Title: Comparing Blood Glucose Control Intraoperative Between Insulin Drip vs. Insulin Boluses Will Provide Valuable Information on the Optimal Method for Achieving Blood Glucose Control Intraoperatively.
Acronym: RANDOM-IB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Mohammed Alrefai, Principal Investigator, King Faisal Specialist Hospital & Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB # 2023-45
Record Dates: First submitted 2025-06-24; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Hypoglycemia (Diabetic)
MeSH Terms: conditions — Hypoglycemia

STUDY DESIGN:
Intervention Model Description: Simple randomization will be used for randomization. The participants will be randomized into two groups based on methods of insulin delivery.
  * Group A: Insulin drip will be administered at a starting rate of 2 units/hour and titrated to maintain blood glucose levels between 80-180 mg/dL.
  * Group B: Insulin boluses will be administered every 30 minutes to maintain blood glucose levels between 80-180 mg/dL.
  Insulin boluses will be considered as a control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Insulin drip (Experimental)
  Interventions: Drug: Insulin Drip Therapy
- Insulin boluses (Other): Control group
  Interventions: Drug: Insulin boluses

INTERVENTIONS:
Drug: Insulin Drip Therapy — Simple randomization will be used for randomization. The participants will be randomized into two groups based on methods of insulin delivery.
  * Group A: Insulin drip will be administered at a starting rate of 2 units/hour and titrated to maintain blood glucose levels between 80-180 mg/dL.
  * Group B: Insulin boluses will be administered every 30 minutes to maintain blood glucose levels between 80-180 mg/dL.
  Insulin boluses will be considered as a control group.
  Arms: Insulin drip
Drug: Insulin boluses — Insulin boluses will be administered every 30 minutes to maintain blood glucose levels between 80-180 mg/dL.
  Insulin boluses will be considered as a control group
  Arms: Insulin boluses

SUMMARY:
Cardiac surgery patients often experience elevated blood glucose levels, which can lead to poor surgical outcomes and increased postoperative complications. Therefore, tight blood glucose control during surgery is important. Currently, there is no consensus on the best method for blood glucose control during cardiac surgery. This proposal aims to perform a randomized controlled trial to compare blood glucose control intraoperatively using an insulin drip versus insulin boluses. The primary objective of the study is to compare blood glucose control intraoperatively between patients who receive insulin drip and patients who receive insulin boluses during adult cardiac surgery. This study will be a randomized controlled trial in which adult patients undergoing cardiac surgery will be randomized into two groups: insulin drip and insulin boluses. Patients with a history of diabetes or those currently taking antidiabetic medications will be included in the study. This randomized controlled trial will provide valuable information on the optimal method for achieving blood glucose control intraoperatively. The results of this study may help improve patient outcomes and reduce the incidence of postoperative complications.

DETAILED DESCRIPTION:
Study Title:

A Randomized Controlled Trial Comparing Intraoperative Blood Glucose Control Between Insulin Drip Versus Insulin Boluses in Adult Cardiac Surgery Patients

Sponsor and Funding:

Sponsor: None

Funding Organization: King Faisal Specialist Hospital & Research Center, Jeddah

Study Site: Single center at King Faisal Specialist Hospital & Research Center, Jeddah

Background and Rationale:

Maintaining optimal blood glucose levels during cardiac surgery is critical for reducing postoperative complications and improving patient outcomes. Current intraoperative glucose management strategies vary, with insulin administered either continuously via infusion (drip) or intermittently as boluses. This trial investigates which method provides superior glucose control intraoperatively.

Study Design:

This is a prospective, single-center, randomized controlled trial (RCT) with two parallel arms:

Insulin drip group (continuous infusion)

Insulin bolus group (intermittent dosing)

Objectives:

Primary Objective: To compare the effectiveness of insulin drip versus insulin boluses in maintaining intraoperative blood glucose within target ranges during adult cardiac surgery.

Secondary Objectives: To assess the incidence of hypoglycemic events, insulin dose adjustments, duration of ICU stay, lactate clearance, and wound infection rates at 7- and 30-days post-surgery.

Endpoints:

Primary Endpoint: Rate of severe hypoglycemia during surgery.

Secondary Endpoints: ICU length of stay, postoperative lactate clearance, incidence of surgical wound infections at 7- and 30-days post-operation.

Participants:

Sample Size: 384 total participants, randomized equally into two groups (192 per group).

Inclusion Criteria: Adults aged over 18 years undergoing cardiac surgery, preoperative blood glucose between 80-180 mg/dL, with a documented history of diabetes.

Exclusion Criteria: Known intolerance to insulin, severe hepatic dysfunction, recent hypoglycemic episodes.

Intervention Protocols:

Insulin Drip Group: Continuous intravenous insulin infusion initiated at 2 units/hour, titrated to maintain target intraoperative glucose levels.

Insulin Bolus Group: Insulin administered as bolus doses every 30 minutes, adjusted based on glucose monitoring.

Data Collection and Follow-up:

Blood glucose and other relevant clinical parameters are monitored intraoperatively. Participants are followed postoperatively at 1 week, 1 month, 6 months, and 1 year to evaluate long-term outcomes and complications. The total anticipated duration of the trial is 4 years.

Statistical Analysis:

Data analysis will involve calculation of relative risk for hypoglycemia and other categorical outcomes. Time-to-event data will be analyzed using log-rank tests. Statistical significance is defined as p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (above 18 y of age undergoing Cardiac surgery with preoperative blood glucose level (80 -180 mg/dL)
* Patient with History of diabetes and those taking antidiabetics medications.

Exclusion Criteria:

* Patients with known allergy or insulin intolerance.
* Patients with severe hepatic Dysfunction.
* Patient with History of hypoglycemic events in the past 6 month prior to surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2029-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Rate of severe hypoglycemia | one year

SECONDARY OUTCOMES:
Duration of ICU stay | 24 hours
The incidence of wound infection | 7-30 days
lactate clearance | From the end of surgery to 6 hours postoperatively
  the percentage decrease in blood lactate concentration

DOCUMENTS (2):
  • Study Protocol (2024-10-10): https://cdn.clinicaltrials.gov/large-docs/88/NCT07056088/Prot_000.pdf
  • Informed Consent Form (2024-11-04): https://cdn.clinicaltrials.gov/large-docs/88/NCT07056088/ICF_001.pdf